CLINICAL TRIAL: NCT00546520
Title: A 3-period Double-blind, Cross-over Study on the Onset of Action of Inhaled Ciclesonide (7 Days of 400 mcg Sid Versus 800 mcg Bid Versus Placebo) on Airway Responsiveness to Adenosine Monophosphate (AMP), Sputum Eosinophiles and Exhaled Breath Nitric Oxide (NO) in Patients With Asthma
Brief Title: Effect of Inhaled Ciclesonide in Adult Patients With Asthma (BY9010/M1-125)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: BY9010/M1-125
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Asthma
Keywords: Asthma; Ciclesonide; Airway hyperresponsiveness; Sputum; Nitric oxide
MeSH Terms: conditions — Asthma; Respiratory Hypersensitivity | interventions — ciclesonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ciclesonide

SUMMARY:
Ciclesonide is a novel inhaled corticosteroid for the treatment of asthma. In this study the effect of ciclesonide on airway hyperresponsiveness (AHR), exhaled nitric oxide (NO), and induced sputum inflammatory biomarkers will be evaluated.

ELIGIBILITY:
Main inclusion criteria:

* Out-patients
* Written informed consent
* History of atopic disease
* History of perennial bronchial asthma for at least 6 months as defined by ATS criteria
* Current use of only inhaled short acting beta-2-agonist as required (for at least 4 weeks prior to baseline period B0)
* Stable asthma, i.e. no exacerbation or relevant respiratory tract infection within 2 months prior to study start
* FEV1 ≥ 70% predicted
* Hyperreactivity to AMP (PC20FEV1 < 25 mg/ml)
* Good health with the exception of asthma
* Non-smokers as well as ex-smokers with either = 10 pack-years or more than 6 months of smoking abstinence

Main exclusion criteria:

* Concomitant severe diseases or diseases which are contraindications for the use of inhaled steroids (e.g. lung tuberculosis)
* Clinically relevant abnormal laboratory values suggesting an unknown disease and requiring further clinical evaluation
* Use of systemic steroids 4 weeks (injectable depot steroids 6 weeks) before entry into the baseline period, or more than 3 times during the last 6 months
* Pregnancy or intention to become pregnant during the course of the study, breast feeding, lack of safe contraception in heterosexually active female patients of child-bearing potential, or postmenopausal for less than one year
* COPD (i.e. chronic bronchitis or emphysema) and/or other relevant lung diseases
* Known or suspected hypersensitivity to inhaled steroids or to the other excipients of the metered dose inhalers
* Immunotherapy within one month prior to B0 and/or during the entire study duration

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2002-04; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
PC20FEV1 (AMP)

SECONDARY OUTCOMES:
Baseline FEV1 from spirometry, exhaled NO, eosinophils, basophils, and mast cells determined from induced sputum; Safety variables: Physical examination, vital signs, ECG, laboratory work-up, and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- "Altana Pharma/Nycomed", London, United Kingdom